CLINICAL TRIAL: NCT01317433
Title: Pre-emptive Cycline Treatment on Cetuximab-induced Skin Toxicity in Patients With Metastatic Colorectal Cancer Treated With an Intensified FOLFIRI.
Brief Title: Pre-emptive Cycline Treatment on Cetuximab Induced Skin Toxicity in Colorectal Cancer
Acronym: SKINUX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study stopped due to a lack of recruitment
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPP-450; 2010-019140-39 (EudraCT Number)
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Colorectal Cancer Metastatic; Skin Toxicity
Keywords: Metastatic Colorectal Cancer; K-RAS wild-type; FOLFIRI; Cetuximab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Doxycycline; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Intensified FOLFIRI plus Cetuximab + Doxycycline 100 mg daily per os to start 7 days before Cetuximab for 6 weeks + skin moisturizers (Dexeryl), sun protection.
  Interventions: Drug: Doxycycline; Drug: Cetuximab
- Arm B (Active Comparator): Intensified FOLFIRI plus Cetuximab + skin moisturizers (Dexeryl), sun protection.
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Doxycycline — Doxycycline 100 mg daily per os to start 7 days before Cetuximab for 6 weeks.
  Arms: Arm A
Drug: Cetuximab — 500 mg/m² IV infusion of 60 minutes every 15 days

SUMMARY:
The aim of this study is to test the role of cycline in the prevention of acne-like skin rash in metastatic colorectal patients treated with Cetuximab and intensified FOLFIRI.

DETAILED DESCRIPTION:
Cetuximab, an Epidermal Growth Factor Receptor (EGFR) inhibitor, has shown to improve FOLFIRI efficacy up to 59.3% OR, in wild KRAS patients with advanced colorectal cancer. Skin toxicity occurs in 81.6% of patients as an acne-like skin rash developed on the face and the trunk inducing pain, decreasing quality of life and drug compliance. Over 104 patients enrolled in a phase II clinical trial sponsored by Center Paul Papin (NCT 00 559741), a grade > or = 2 cetuximab-acneiform rash occured in 51 patients (49%). In this trial Cetuximab was combined with a FOLFIRI intensified (5-FU intensification based on pharmacokinetics and pharmacogenetic studies of UGT1A1 status and DPD). Until now, no pre-emptive skin toxicity treatment with cycline has been demonstrated. Because of cycline's anti inflammatory properties and their use in inflammatory acne, cycline could prevent cetuximab-induced skin rash. In a randomized double-blind placebo-controlled phase III trial, Jatoi et al., failed to highlight any cycline effect on 61 patients. On the other hand, the STEPP study (95 pts) showed the impact of cycline to prevent panitumumab related skin toxicities. Our primary objective is to reduce the incidence of grade > or = 2 acne-like skin rash by 30% with a 6 weeks pre-emptive cycline treatment in patients with metastatic colorectal cancer undergoing cetuximab therapy.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic colorectal cancer, histologically confirmed, first or second metastatic line
* K-RAS wild-type
* Adjuvant prior chemotherapy allowed provided that all toxicities are grade < or = 1 (excepted alopecia and neuropathy)
* Age between 18 and 80 years
* WHO Performance Status < or = 2
* Complete initial assessment before first treatment administration for imaging and pharmacogenetic, within 15 days for biology, and within 7 days for clinical examination.
* Haematologic and hepatic parameters : neutrophils > or = 1500 /mm3, platelets > or = 100000/mm3, Total bilirubin < or 2 x ULN, AST and ALT < or = 3 x ULN, APL < or = 5 x ULN
* Absence of total dihydropyrimidine dehydrogenase deficiency
* Patient able to comply with study requirements
* Signed written informed consent

Exclusion Criteria:

* History or presence of an other cancer, excepted cutaneous cancer (basocellular carcinoma), in situ cancer of the cervix or breast cancer curatively treated
* Any other concomitant anti-cancer therapy
* Prior anti EGFR therapy, anti angiogenic therapy is allowed
* Prior cyclines hypersensitivity
* Treatment with cyclines within 7 days before randomization
* Presence of a rash at randomization time
* Symptomatic or uncontrolled ventral nervous system metastases
* Total dihydropyrimidine dehydrogenase deficiency
* No recovery of any toxicity Grade < or = 1 related to a past anticancerous treatment excepted for alopecia and neuropathy
* Active inflammatory bowel disease or other bowel
* Significant serious pathology or any unstable medical condition (cardiac pathology uncontrolled, myocardial infarction within 6 months before enrollment, systemic active uncontrolled infection)
* atropine contra-indication
* any investigational agent without marketing authorization within 4 weeks before enrollment
* Patient who is pregnant or breast feeding
* Woman or man of childbearing potential not consenting to use adequate contraceptive precautions during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-12-29 (Actual); Primary Completion 2016-10-10 (Actual); Study Completion 2016-10-10 (Actual)

PRIMARY OUTCOMES:
reduction of Grade > or = 2 acne-like skin rash by 30% | 6 weeks of pre-emptive cycline treatment
  Skin tolerance will be assessed by a dermatologist at each cycle and NCI CTCAE v4.0 will be use for grading. Skin standardized photographs will be done at every cycle and a central double blind review wil be planned. Time to first occurence of grade > or =2 skin toxicity will be assessed, and specificity.

SECONDARY OUTCOMES:
skin tolerance assessment | Until the end of Cetuximab treatment
  Skin tolerance will be assessed weekly by a dermatologist from C1 to C3, and biweekly from C4 to C6 and NCI CTCAE v4.0 will be use for grading. All grade > or = 1 skin and hair/nails toxicities will be reported. Time to most severe skin toxicity will be assessed. Quality of life questionnaires with a skin interest (DLQI) will be evaluated at baseline and at each cycle.
Non skin toxicities assessment | Until the end of chemotherapy treatment
  For non skin toxicities, only grade > or = 3 will be reported.
Efficacy Objective Response (OR) assessment | Until the end of chemotherapy treatment
  Efficacy OR (Complete Response + Partial Response) will be assessed by the investigator with usual tumoral evaluation. Tumoral evaluation will be assessed with the same exam throughout the trial.
Biological correlation with response and survival | 3 years
  Biological correlation with response and survival will be tested for KRAS, BRAF, PI3K,PTEN, epiregulin, amphiregulin, IGF1, Syndecan-1, UBE2C, EGFR polymorphism.
Time To Progression and Overall Survival | 3 years
Resectability rate | Until the end of chemotherapy treatment

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Capitain, MD, PhD, Principal Investigator — Institut Cancerologie de l'Ouest
Locations (5):
- France (5):
  - ICO Paul Papin, Angers
  - CHU Jean Minjoz, Besançon
  - CHU Morvan, Brest
  - Centre Hospitalier, Cholet
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon